CLINICAL TRIAL: NCT01113216
Title: Genetic Modifiers of Cystic Fibrosis Related Diabetes
Status: Enrolling by invitation | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Cystic Fibrosis Foundation (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Minnesota (Other); Northwestern University (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00005921; K23DK083551 (NIH); CFF-CFRD01 (Other: Other)
Record Dates: First submitted 2010-04-28; First posted 2010-04-29 (Estimated); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Cystic Fibrosis Related Diabetes
Keywords: CF; CFRD; Diabetes; Genetic Modifiers
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be drawn from study participants and their parents. Two tablespoons of blood (one tablespoon in small children) will be drawn by standard techniques from a vein in the arm. Whenever possible, blood samples for this study will be collected at the same time that it is done for medically needed blood tests. This blood will be used to extract DNA and to establish cell lines that we will store as a permanent source of DNA. We will compare your clinical symptoms with your DNA to see if additional genes that affect CF symptoms can be found. Some serum and plasma will be stored for later testing, as additional knowledge becomes available. Any tests done in the future with your stored blood samples or your DNA will only be to answer questions about genes for CF.
Oversight: Data Monitoring Committee: No

SUMMARY:
This research is being done to find the genes and other factors that are responsible for differences among persons with cystic fibrosis. We are particularly interested in the factors that relate to the development of Cystic Fibrosis Related Diabetes (CFRD).

DETAILED DESCRIPTION:
The study is recruiting people with cystic fibrosis (CF). The medical record is being extracted, and a blood sample is taken for DNA. The DNA samples are tested for variation both at the cystic fibrosis transmembrane conductance regulator (CFTR) gene (the CF gene) and over the entire rest of the genome. Using large numbers of people with CF, and knowing who does and does not have CFRD, we identify genetic variations that associate with CFRD. Knowing these variations allows us to better understand the causes of CFRD, and with enough information, better to predict CFRD and identify people at particularly high or low risk of CFRD. People participating in this study also have the option to participate in related studies of other metabolic traits in CF such as over- and underweight.

ELIGIBILITY:
Inclusion Criteria:

* Any person with Cystic Fibrosis and his/her parents.

Exclusion Criteria:

* None

Ages: 3 Months to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals affected with Cystic Fibrosis and family members
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2008-04; Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Identification of Genes or other factors that influence the development of CFRD | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Blackman, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - Children's Memorial Hospital, Chicago, Illinois
  - Johns Hopkins Medicine, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aksit MA, Pace RG, Vecchio-Pagan B, Ling H, Rommens JM, Boelle PY, Guillot L, Raraigh KS, Pugh E, Zhang P, Strug LJ, Drumm ML, Knowles MR, Cutting GR, Corvol H, Blackman SM. Genetic Modifiers of Cystic Fibrosis-Related Diabetes Have Extensive Overlap With Type 2 Diabetes and Related Traits. J Clin Endocrinol Metab. 2020 May 1;105(5):1401-15. doi: 10.1210/clinem/dgz102. PMID 31697830
- [Background] Aksit MA, Ling H, Pace RG, Raraigh KS, Onchiri F, Faino AV, Pagel K, Pugh E, Stilp AM, Sun Q, Blue EE, Wright FA, Zhou YH, Bamshad MJ, Gibson RL, Knowles MR, Cutting GR, Blackman SM; CF Genome Project. Pleiotropic modifiers of age-related diabetes and neonatal intestinal obstruction in cystic fibrosis. Am J Hum Genet. 2022 Oct 6;109(10):1894-1908. doi: 10.1016/j.ajhg.2022.09.004. PMID 36206743
- [Result] Blackman SM, Hsu S, Vanscoy LL, Collaco JM, Ritter SE, Naughton K, Cutting GR. Genetic modifiers play a substantial role in diabetes complicating cystic fibrosis. J Clin Endocrinol Metab. 2009 Apr;94(4):1302-9. doi: 10.1210/jc.2008-2186. Epub 2009 Jan 6. PMID 19126627
- [Result] Blackman SM, Hsu S, Ritter SE, Naughton KM, Wright FA, Drumm ML, Knowles MR, Cutting GR. A susceptibility gene for type 2 diabetes confers substantial risk for diabetes complicating cystic fibrosis. Diabetologia. 2009 Sep;52(9):1858-65. doi: 10.1007/s00125-009-1436-2. Epub 2009 Jul 8. PMID 19585101
- [Result] Blackman SM, Commander CW, Watson C, Arcara KM, Strug LJ, Stonebraker JR, Wright FA, Rommens JM, Sun L, Pace RG, Norris SA, Durie PR, Drumm ML, Knowles MR, Cutting GR. Genetic modifiers of cystic fibrosis-related diabetes. Diabetes. 2013 Oct;62(10):3627-35. doi: 10.2337/db13-0510. Epub 2013 May 13. PMID 23670970